CLINICAL TRIAL: NCT05596773
Title: Community-Based Chronic Disease Care in Rural Lesotho: The ComBaCaL Cohort Study
Brief Title: Community-Based Chronic Disease Care in Rural Lesotho
Acronym: ComBaCaL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Agency for Development and Cooperation (SDC) (Unknown); World Diabetes Foundation (WDF) (Unknown); SolidarMed (Other)
Responsible Party: Sponsor
Other Study IDs: AO_2022-00058; ex21Labhardt
Record Dates: First submitted 2022-10-12; First posted 2022-10-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Non-communicable Diseases (NCDs)
Keywords: Community-Based Chronic Disease Care Lesotho (ComBaCaL); Chronic Care Village Health Worker (CC-VHWs); eHealth application (ComBaCaL app); Lesotho; low- and middle-income countries (LMICs); Arterial hypertension (aHT); Diabetes mellitus (DM)
MeSH Terms: conditions — Noncommunicable Diseases; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma or dried blood spot samples of cohort participants may be collected for storage and future analysis. No human genome analysis will be conducted on the samples collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This ComBaCaL cohort study is to assess the impact of community-based, lay-led chronic disease screening and care interventions in rural Lesotho. It aims to establish a prospective research and service delivery platform in rural Lesotho that is managed by eHealth-supported Chronic Care Village Health Worker (CC-VHWs) providing regular chronic disease screening, monitoring and referral services. The implementation outcomes of the cohort as well as the effect of the cohort activities on disease-specific care cascades will be assessed. Subsequently, nested trials to assess the effectiveness of specific chronic disease control interventions will be developed. Measurements and data entry will be conducted by CC-VHWs. The CC-VHWs will be equipped with the essential tools required for chronic disease monitoring in the community (i.e. BP machines, scales, measuring band, glucometers, and urine dipsticks). They will undergo a theoretical and practical training covering all aspects required for correct data collection and chronic disease screening, diagnosing, referral and counselling services. At every visit, the CC-VHW will screen participants for warning signs and symptoms (i.e. shortness of breath, severe headache, chest pain, new-onset confusion, impaired consciousness, severely impaired general state of health) and refer participants to the closest health centre in case of any danger-sign. The CC-VHWs will be continuously monitored and supervised by health centre nurses of the respective village's catchment area, mainly through direct interaction during monthly VHW meetings and by CC nurses through field visits, remote interaction via phone calls or messages sent via the ComBaCaL app and through direct contact during the monthly VHW meetings at the health centre. The CC-VHWs are embedded within the Lesotho MoH VHW program and may during the project period be trained and equipped to provide further routine services in their communities.

DETAILED DESCRIPTION:
Globally, non-communicable diseases (NCDs) are the leading cause of death and disability with a particularly high burden in Low- and middle-income countries (LMICs), where more than 75% of all premature NCD deaths occur. Lesotho is a typical example of an African LMIC where NCDs are overtaking Human immunodeficiency virus (HIV)/AIDS and other infectious diseases as major cause of disability, morbidity and early death. HIV and NCDs are chronic diseases and share several characteristics such as the asymptomatic initial phase, progression to complications with disability and early death, and need for life-long treatment. The Ministry of Health (MoH) of Lesotho has therefore proposed in its NCD strategic plan that lessons learnt from the HIV program should be taken up to similarly reduce the existing access barriers to NCD care. Two scoping reviews have shown that the evidence on how and to what extent task shifting to lay workers can successfully be implemented for NCDs in sub-Sahara Africa is very limited. This open, prospective cohort study aims at generating evidence on community-based screening, diagnosis and management of uncomplicated arterial hypertension (aHT), Diabetes mellitus (DM) and other chronic diseases by lay Village health worker (VHWs) in a rural sub-Saharan African setting. It is to establish an observational cohort (ComBaCaL cohort) with regular monitoring of chronic disease indicators and risk factors in Butha-Buthe and Mokhothlong districts in Lesotho that will be managed by lay Chronic Care Village Health Workers (CC-VHWs), supported by a dedicated tablet-based eHealth application. The prevalence of common chronic diseases and associated risk factors in the cohort population and will be assessed and their development over time will be monitored. Initial focus will be on aHT, DM, cardiovascular disease risk factors (CVDRFs) and HIV. Other conditions may be included at a later stage. The effect of the ComBaCaL activities on condition- specific care cascade outcomes, such as screening coverage, disease awareness, linkage to care, engagement in care and disease control rates will be analyzed. Cohort variables will be assessed at baseline and pre-specified analyses to assess the effect of the ComBaCaL on chronic disease care cascades will be conducted at six months (range 150-240 days) and twelve months (range 300-480 days) after enrolment. Variables which may change over time will be reassessed during follow-up visits at intervals of around six months.

The ComBaCaL cohort will be a platform for nested pragmatic trials (Trials within a Cohort, TwiCs) assessing chronic disease care interventions.

ELIGIBILITY:
Inclusion Criteria village level:

* Village size of 40 to 100 households
* Village consent obtained from village chief
* Possibility to identify or recruit a CC-VHW from the village population meeting the following requirements which are largely in line with the criteria of the Lesotho VHW Program Policy:

  o Criteria of the Lesotho Village Health Program Policy:
* Having primary residence in the village (according to village chief)
* Having a proven record of trustworthiness in the resident village
* Having proven ability to maintain confidentiality on public matters
* Being aged between 20 and 50 years
* Being able to provide written reports and being able to do basic mathematical calculations
* Having at least educational level equivalent to high school leaving certificate (Junior Certificate)

  o Additional ComBaCaL criteria:
* Having the ability and willingness to work with a tablet-based eHealth tool
* Having good social and communication skills
* Having the ability and willingness to interact with health professionals and the village population
* Being able to speak, understand and write in English-
* Having successfully completed the ComBaCaL CC-VHW training including final assessment

Inclusion criteria individual level:

* Having primary residence in the village (self-reported at time of enrolment)
* Being able and willing to consent to participation or in case of individuals aged below 18

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inhabitants of around 100 (range 90-110) randomly selected villages in rural Lesotho. The estimated mean number of inhabitants per village is 200. All inhabitants will be approached for consent and all consenting individuals (assent plus guardian consent for adolescents (10-17 years), guardian consent for children <10 years) will be enrolled into the ComBaCaL cohort.
Sampling Method: Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Screening coverage | At baseline
  Screening coverage for aHT and (pre)DM, defined as the proportion of screening-eligible participants that have been screened for the respective disease within the previous 3 years
Disease awareness | At baseline
  Disease awareness for aHT and (pre)DM, defined as the proportion of participants diagnosed with aHT or (pre)DM that are aware of their condition
Linkage to care | Up to 3 years after enrolment
  Linkage to care for aHT and DM, defined as the number of participants with aHT or (pre)DM who (re)started drug treatment for their respective condition since enrolment
Engagement in care | Up to 3 years after enrolment
  Engagement in care for aHT and DM, defined as the number of participants with aHT or (pre)DM who had a check-up measurement (BG or HbA1C for (pre)DM, BP for aHT) or drug refill within the last 180 days for their condition
Disease control level | Up to 3 years after enrolment
  Disease control level for aHT and DM, defined as the number of participants with aHT or DM who are reaching disease-specific treatment targets (BP <140/90 mmHg for aHT, fasting blood glucose (FBG) < 7mmol/l and/or HbA1C <7.0% for DM)
Occurrence of clinically relevant events (number) | Up to 3 years after enrolment
  Occurrence of clinically relevant events (Clinical event of special interest (CESI), Serious clinical event (SCE), Serious clinical event of special interest (SCESI), as defined by the protocol

OTHER OUTCOMES:
Feasibility of ComBaCaL's communitybased chronic disease care activities among participants, CC-VHWs and involved healthcare professionals using mixed-methods assessments | Up to 3 years
Acceptability of ComBaCaL's communitybased chronic disease care activities among participants, CC-VHWs and involved healthcare professionals using mixed-methods assessments | Up to 3 years
Satisfaction of ComBaCaL's communitybased chronic disease care activities among participants, CC-VHWs and involved healthcare professionals using mixed-methods assessments | Up to 3 years
Perceived appropriateness of ComBaCaL's communitybased chronic disease care activities among participants, CC-VHWs and involved healthcare professionals using mixed-methods assessments | Up to 3 years
Number of households visited by CC-VHW | Up to 3 years
Number of individuals monitored by one CC-VHW | Up to 3 years
Number of individuals newly diagnosed with a chronic condition | Up to 3 years
Number of villages inhabitants refusing community-based chronic disease screening or referral to health facility for further management after diagnosis | Up to 3 years
Resource use of the ComBaCaL activities, including time-and-motion studies among CCVHWs | Up to 3 years
Cost of the ComBaCaL activities, including time-and-motion studies among CCVHWs | Up to 3 years
Completeness of the data collected by CC-VHWs | Up to 3 years
Adherence to clinical algorithms provided via the eHealth application | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, Prof. Dr. med., Principal Investigator — Division of Clinical Epidemiology, University Hospital Basel, University of Basel; Alain Amstutz, MD, Principal Investigator — Division of Clinical Epidemiology, University Hospital Basel, University of Basel
Locations (2):
- Solidarmed Lesotho, Maseru, Lesotho
- Division of Clinical Epidemiology, University Hospital Basel, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
• An anonymized key dataset will be made freely available in an appropriate repository, such as zenodo.org, alongside the publication of study results. Besides removal of variables not required for key analysis, we will remove participant identifier, study site and exact date information. Requests for access to more detailed data may be made to the corresponding author by submitting a proposal, which will be reviewed by the trial consortium.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: • Within 3 months after publication of primary results
Access Criteria: • Open access

REFERENCES:
- [Derived] Gerber F, Sanchez-Samaniego G, Tahirsylaj T, Lejone TI, Lee T, Raeber F, Chitja M, Mathulise M, Kabi T, Mokaeane M, Maphenchane M, Molulela M, Mota M, Masike S, Bane M, Makabateng R, Khomolishoele M, Sematle M, Gupta R, Ayakaka I, Sao L, Tlahali M, Phaaroe S, Litaba M, Mphunyane M, Basler DB, Kindler K, Grimm P, Seelig E, Burkard T, Briel M, Chammartin F, Amstutz A, Labhardt ND. Cohort profile: the open, prospective Community-Based chronic Care Lesotho (ComBaCaL) cohort - design, baseline chronic disease risk factors and hypertension and diabetes care cascades. BMJ Open. 2025 Jul 25;15(7):e093852. doi: 10.1136/bmjopen-2024-093852. PMID 40713039

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05596773/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05596773/ICF_001.pdf